CLINICAL TRIAL: NCT02552875
Title: Shortening of the Twitch Stabilization Period by Tetanic Stimulation in Acceleromyography in Children and Young Adults
Acronym: STSTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Christoph Unterbuchner, Dr. med. Christoph Unterbuchner, DESA, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-101-0114
Record Dates: First submitted 2014-07-29; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Train-of-Four-Monitoring
Keywords: Acceleromyography; staircase phenomenon; tetanic stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetanic Stimulation (Active Comparator): 50 Hz tetanic stimulation for 5 seconds before TOF-twitch stabilization at the one arm
  Interventions: Other: Tetanic stimulation
- Staircase Stimulation (Active Comparator): TOF-twitch stabilisation without 50 Hz tetanic stimulation at the contralateral arm
  Interventions: Other: Staircase Stimulation

INTERVENTIONS:
Other: Tetanic stimulation — 50 Hz tetanic stimulation before TOF-twitch stabilization with the aim to eliminate the staircase phenomenon
  Arms: Tetanic Stimulation
Other: Staircase Stimulation — TOF-twitch stabilization without 50 Hz tetanic stimulation with the aim to verify the staircase phenomenon
  Arms: Staircase Stimulation

SUMMARY:
Repetitive nerve stimulation is used to monitor the neuromuscular transmission function in infants, children and adults after the application of muscle relaxants. During repetitive stimulation of a motor nerve, amplitude of contractions of the corresponding muscle will increase to a plateau (twitch potentiation), which is known as the staircase phenomenon.

There is no systematic information about the staircase phenomenon of the adductor pollices muscle (ulnar nerve) in children between 1 month and 18 years .

In adults , a 50-Hz tetanus administered before initial twitch stabilization is able to shorten the twitch stabilization period and to eliminate this staircase phenomenon.

The purpose of this study is to investigate the characteristics of twitch potentiation in children between 1 month and 18 years by using acceleromyography.

In addition we investigate whether application of a 50-Hz tetanic stimulation is able to eliminate the twitch potentiation like in adults.

DETAILED DESCRIPTION:
1. Background:

   Acceleromyography at the adductor pollices muscle (ulnar nerve stimulation) is used to monitor the neuromuscular transmission function in infants, children and adults after the application of muscle relaxants. During repetitive stimulation of a motor nerve, amplitude of contractions of the corresponding muscle will increase to a plateau (twitch potentiation), which is known as the staircase phenomenon. This effect may influence the onset time and duration of twitch depression after the application of muscle relaxants. The staircase effect during the baseline stabilization period presents in a shorter time course and at lower degrees in smaller infants. In older infants, staircase effect presents in a longer period and is able to influence duration of twitch depression after the administration of muscle relaxants.

   There is no information about the staircase phenomenon at the adductor pollices muscle (ulnar nerve stimulation) in children between 1 month and 21 years.

   In adults , a 50-Hz tetanus administered before initial twitch stabilization is able to shorten the twitch stabilization period and to eliminate this phenomenon.
2. Aim of the study:

   The purpose of this controlled, randomised, pragmatic study is to investigate the characteristics of twitch potentiation (T1%, first twitch of TOF-stimulation; TOFR, Train-of-Four-ratio) in children between 1 month and 21 years by using acceleromyography. In addition we stimulate the right and the left arm simultaneously with acceleromyography (TOF-stimulation). At the one hand a 50 Hz tetanus will be administered before twitch stabilization (TOF-stimulation). At the other hand TOF-stimulation for twitch stabilization will be started without tetanic stimulation
3. Methods:

   Anaesthesia will be induced and maintained without muscle relaxants by propofol and remifentanil. After this acceleromyography will be performed simultaneously at the right and the left arm (adductor pollices muscle, ulnar nerve). At the one hand a 50 Hz tetanus will be administered before twitch stabilization (TOF-stimulation). At the contralateral side TOF-stimulation for twitch stabilization will be started without tetanus. TOF measurements will be collected by 2 TOF Watch SX and two notebooks for the course of 30 minutes.
4. Inclusion criterions/ groups

   -general anesthesia (total intravenous anaesthesia)

   Groups (total amount= 80)
   * group A: 18-21 years; n= 10
   * group B: 12-18 years; n= 10
   * group C: 6-12 years; n= 10
   * group D: 3-6 years; n= 10
   * group E: 25-60 months; n= 10
   * group F: 12-24 months; n= 10
   * group G: 6-11 months; n= 10
   * group H: 1-5 months; n= 10.
5. Exclusion criterions

   * participation in another trial
   * refusal of participation
   * state after burns
   * diabetes mellitus
   * reflux disease
   * difficult airway
   * pregnancy

Medications:

* volatile anesthetics
* antibiotics (aminoglycosides, polymyxin, clindamycin, lincomycin, tetracyclines)
* local anesthetics
* magnesium
* lithium
* Ca-chanel-blockers
* furosemide
* theophylline
* phenytoin
* cyclophosphamide
* metoclopramide
* β-blockers

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia

Exclusion Criteria:

* participation in another trial
* refusal of participation
* state after burns
* diabetes mellitus
* reflux disease
* difficult airway
* pregnancy

Medications:

* volatile anesthetics
* antibiotics (Aminoglykoside, Polymyxin, Clindamycin, Lincomycin, Tetrazykline)
* local anesthetics
* magnesium
* Litium
* Ca-chanel-blockers
* furosemid
* theophyllin
* phenytoin
* cyclophosphamide
* metoclopramide
* β-blockers

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
T1% measurement | 30 minutes
  T1% increase dependent on stimulation with and without a 50 Hz tetanic stimulation

SECONDARY OUTCOMES:
TOFR% maesurement | 30 minutes
  TOFR%course dependent on stimulation with and without a 50 Hz tetanic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Unterbuchner, MD, Principal Investigator — University Medical Center Regensburg, Germany
Locations (1):
- University Medical Center Regensburg, Department of Anaesthesiology, Regensburg, Germany

REFERENCES:
- [Background] Saldien V, Vermeyen KM. Neuromuscular transmission monitoring in children. Paediatr Anaesth. 2004 Apr;14(4):289-92. doi: 10.1046/j.1460-9592.2003.01152.x. No abstract available. PMID 15078372
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Lee GC, Iyengar S, Szenohradszky J, Caldwell JE, Wright PM, Brown R, Lau M, Luks A, Fisher DM. Improving the design of muscle relaxant studies. Stabilization period and tetanic recruitment. Anesthesiology. 1997 Jan;86(1):48-54. doi: 10.1097/00000542-199701000-00008. PMID 9009939
- [Background] Zhou ZJ, Wang X, Zheng S, Zhang XF. The characteristics of the staircase phenomenon during the period of twitch stabilization in infants in TOF mode. Paediatr Anaesth. 2013 Apr;23(4):322-7. doi: 10.1111/pan.12041. Epub 2012 Oct 17. PMID 23072260
- [Background] Kopman AF, Kumar S, Klewicka MM, Neuman GG. The staircase phenomenon: implications for monitoring of neuromuscular transmission. Anesthesiology. 2001 Aug;95(2):403-7. doi: 10.1097/00000542-200108000-00023. PMID 11506113
- [Background] Driessen JJ, Robertson EN, Booij LH. Acceleromyography in neonates and small infants: baseline calibration and recovery of the responses after neuromuscular blockade with rocuronium. Eur J Anaesthesiol. 2005 Jan;22(1):11-5. doi: 10.1017/s0265021505000037. PMID 15816566
- [Background] Goudsouzian NG, Standaert FG. The infant and the myoneural junction. Anesth Analg. 1986 Nov;65(11):1208-17. No abstract available. PMID 3532867
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Derived] Unterbuchner C, Werkmann M, Ziegleder R, Kraus S, Seyfried T, Graf B, Zeman F, Blobner M, Sinner B, Metterlein T. Shortening of the twitch stabilization period by tetanic stimulation in acceleromyography in infants, children and young adults (STSTS-Study): a prospective randomised, controlled trial. J Clin Monit Comput. 2020 Dec;34(6):1343-1349. doi: 10.1007/s10877-019-00435-4. Epub 2019 Nov 30. PMID 31786715